CLINICAL TRIAL: NCT05025254
Title: Deep Cognitive Endophenotyping of Parkinson's Disease: A Platform Development and Pilot Study
Brief Title: Cognitive Testing Online in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: McGill University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-6045
Record Dates: First submitted 2021-08-13; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD patients: This is an observational study. The PD patient group will consist of participants who self-report that they have a diagnosis of Parkinson's disease
  Interventions: Other: Neurocognitive testing
- Healthy controls: This is an observational study. The healthy control group will consist of participants who self-report that they do not have a diagnosis of Parkinson's disease
  Interventions: Other: Neurocognitive testing

INTERVENTIONS:
Other: Neurocognitive testing — We are assessing several cognitive domains and have made minor adaptations (reducing the total number of trials or lengthening response windows) to several standard neuropsychology tests including measures of executive function, working memory, visuospatial function, declarative memory, reward processing, response inhibition.
  Overall, the tests we use follow a standard set-up: participants are shown stimuli on the screen and are asked to provide a response using either a keyboard or a mouse, based on a specific set of instructions. We always provide a detailed set of on-screen instructions and a practice phase. In some cases, information about performance is provided in the form of points, in other cases, none is provided.

SUMMARY:
This is a feasibility and pilot study. Though large-scale online neurocognitive testing is increasingly being done in psychiatry, there are no such efforts in Parkinson's research. Thus a large part of this pilot study will be to demonstrate feasibility and reliability, and use this experience to develop a feasible protocol for ongoing research. The specific short-term objectives are:

1. To establish the feasibility of performing large-scale deep cognitive phenotyping using online cognitive testing.
2. To demonstrate that online neurocognitive testing is valid and reliable in a smaller sample of locally recruited participants tested both in-lab and online.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's disease by neurologist or healthy individual with no diagnosis of any neurological illness

Exclusion Criteria:

* Psychotic spectrum disorders, active uncontrolled depression, advanced dementia (i.e. needing assistance with daily activities such as dressing or bathing), major stroke, major head injury, epilepsy requiring anti-seizure medications

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with and without Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Completion rate of cognitive test set (feasibility) | Measured once, as this is a cross-sectional study (time to complete cognitive tests is estimated to be 1.5 hours)
  Proportion of registered participants who complete all the cognitive testing.

SECONDARY OUTCOMES:
Reliability of web-based vs in-person working memory testing (n-back test) | Web-based and in-person testing will occur at two separate time points, at least 1 month apart and no more than 3 months apart
  Intraclass correlation coefficient for web-based vs. in-person performance on the n-back test will be computed
Reliability of web-based vs in-person executive function testing (Stroop test performance) | Web-based and in-person testing will occur at two separate time points, at least 1 month apart and no more than 3 months apart
  Intraclass correlation coefficient for web-based vs. in-person performance on the Stroop test will be computed
Reliability of web-based vs in-person visuospatial function testing (Trail making test performance) | Web-based and in-person testing will occur at two separate time points, at least 1 month apart and no more than 3 months apart
  Intraclass correlation coefficient for web-based vs. in-person performance on the Trail making test will be computed
Reliability of web-based vs in-person declarative memory testing (recognition memory) | Web-based and in-person testing will occur at two separate time points, at least 1 month apart and no more than 3 months apart
  Intraclass correlation coefficient for web-based vs. in-person performance on the image recognition test will be computed
Reliability of web-based vs in-person reward processing testing | Web-based and in-person testing will occur at two separate time points, at least 1 month apart and no more than 3 months apart
  Intraclass correlation coefficient for web-based vs. in-person performance on the probabilistic reward task will be computed

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Sharp, MD, Principal Investigator — McGill University
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada